CLINICAL TRIAL: NCT05126771
Title: Using CUSUM to Analyze the Learning Curve of Aortic Arch Replacement Surgery in Chinese Mainland With Stanford Type A Aortic Dissection
Brief Title: Learning Curve of Aortic Arch Replacement Surgery in Chinese Mainland With Stanford Type A Aortic Dissection
Status: Completed | Type: Observational
Sponsor: Yunlong Fan (Other)
Responsible Party: Sponsor-Investigator, Yunlong Fan, Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: chinaPLAGH-66936549
Record Dates: First submitted 2021-11-06; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Cumulative Sum Learning Curves; Stanford Type A Aorta Dissection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
stanford type A aortic dissection is the most common cause of death caused by aortic disease in Chinese mainland. Patients who are hospitalized need immediate surgical treatment.Emergency aortic arch replacement is difficult and risky. Different surgical methods have different effects on postoperative prognosis. Aortic arch replacement is divided into total-arch replacement (Sun's operation) and hemi-arch replacement. In this study, and the learning Curve of Aortic Arch Replacement Surgery was evaluated with cumulative cum curve.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years who underwent surgery for stanford type A aorta dissection without concurrent cardiac Surgery

Exclusion Criteria:

* data miss greater than 10%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age between 18 years and 65 years who underwent standford type A aorta dissection
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary bypass (CPB) time | Intra-operative
  Cardiopulmonary bypass (CPB) time was used as the main variables for evaluation and visualization of the aorta dissection surgery learning curve using Cumulative sum.Cumulative sum (CUSUM) is a statistical method that focuses on results rather than on the process of performing a program skills, it generates graphs that allow for quick detection of deviations from pre-established standards and is an alternative tool that can be used to evaluate the performance of individual program. CUSUM can be generated based on set acceptable and unacceptable failure rates and the degree to which type 1(α) and type 2(β) errors (false positive and false negative errors) will be tolerated. CUSUM was defined as Sn = ∑(Xi -p0), where Xi = 0 for success and Xi = 1 for failure, p0 is the target reference.
Aortic clamping (AC) time | Intra-operative
  Aortic clamping (AC) time was used as the main variables for evaluation and visualization of the aorta dissection surgery learning curve using Cumulative sum.Cumulative sum (CUSUM) is a statistical method that focuses on results rather than on the process of performing a program skills, it generates graphs that allow for quick detection of deviations from pre-established standards and is an alternative tool that can be used to evaluate the performance of individual program. CUSUM can be generated based on set acceptable and unacceptable failure rates and the degree to which type 1(α) and type 2(β) errors (false positive and false negative errors) will be tolerated. CUSUM was defined as Sn = ∑(Xi -p0), where Xi = 0 for success and Xi = 1 for failure, p0 is the target reference.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided